CLINICAL TRIAL: NCT00124293
Title: A Multi Centre Observational Study to Evaluate the Incidence and Magnitude of Haemorrhagic Progression of Cerebral Contusions and the Identification of Important Safety Issues Following Traumatic Brain Injury
Brief Title: Incidence/Magnitude-Haemorrhagic Progression-Cerebral Contusions and Identification (ID) of Safety Issues After Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7CBI-1587
Record Dates: First submitted 2005-06-30; First posted 2005-07-27 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Acquired Bleeding Disorder; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Factor VII
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This study is conducted in North America. The purpose of this study is to evaluate the occurrence and severity of bleeding in brain injury and to identify important safety issues following traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years - 85 Years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were selected from a speciality practice group (Neurosurgery practices with a focus on head trauma. Subjects will have had a mild-to-moderate head injury and require hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2004-10-06 (Actual); Primary Completion 2005-11-23 (Actual); Study Completion 2005-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States
- Novo Nordisk Investigational Site, Mississauga, Canada

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com